CLINICAL TRIAL: NCT01530022
Title: A Multicenter, Randomized, Double-blind, Double-dummy, 2-period Crossover Study of Neuropsychological Effects of Lacosamide and Carbamazepine Immediate Release in Healthy Subjects
Brief Title: Crossover Study of Neuropsychological Effects of Lacosamide and Carbamazepine Immediate Release in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: SP0998
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
Keywords: Lacosamide; Vimpat; Cognition; Mental Processes; Adverse Effects
MeSH Terms: interventions — Lacosamide; Carbamazepine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCM 300 mg/CBZ-IR 600 mg (Other): Crossover sequence of experimental treatment and active comparator
  Interventions: Drug: Lacosamide (LCM); Drug: Carbamazepine Immediate Release (CBZ-IR)
- CBZ-IR 600 mg/LCM 300 mg (Other): Crossover sequence of active comparator and experimental treatment
  Interventions: Drug: Lacosamide (LCM); Drug: Carbamazepine Immediate Release (CBZ-IR)

INTERVENTIONS:
Drug: Lacosamide (LCM) — LCM 300 mg:
  LCM 50 mg and LCM 100 mg white, film-coated oral tablets and Carbamazepine Immediate Release (CBZ-IR) matching placebo capsules.
  Two times daily (morning and evening) during the first 2 weeks of each Titration Period and during the Taper Phases.
  Three times daily (morning, mid-day, and evening) during last week of each Titration Period and 3-week Treatment Period
  Other Names: Vimpat
Drug: Carbamazepine Immediate Release (CBZ-IR) — CBZ-IR 600 mg:
  CBZ-IR 200 mg oral tablets over-encapsulated to double-blind capsules with an overfill.
  LCM matching placebo tablets two times daily (morning and evening) during the first 2 weeks of each Titration Period and during the Taper Phases.
  Three times daily (morning, mid-day, and evening) during last week of each Titration Period and 3-week Treatment Period.
  Other Names: Tegretol IR

SUMMARY:
The primary objective of this Phase 1 crossover study is to evaluate the neuropsychological effects of Lacosamide (LCM) compared to Carbamazepine Immediate Release (CBZ-IR) after administration in healthy subjects. Safety, tolerability, and pharmacokinetic data will also be collected.

DETAILED DESCRIPTION:
Approximately 50 subjects at multiple sites will crossover to receive both treatments (lacosamide [LCM]and carbamazepine immediate release [CBZ-IR]) in a randomized order during the 2 study treatment periods (Treatment Period 1 and Treatment Period 2).

A Screening Visit will be conducted to evaluate subject eligibility for enrollment into the study. Eligible subjects will return up to 21 days after the Screening Visit and begin Treatment Period 1. During Visit 2, eligible subjects will be randomized to receive either LCM 300 mg/day or CBZ-IR 600 mg/day. Subjects will be treated with their first randomized Antiepileptic Drug (AED) for 6 weeks (Titration Period [21 days] and Maintenance Period [21 days]). Subjects then complete a 28-day Taper/Washout Period, during which their first AED will be tapered over 4 days followed by a 24-day Washout Period, where subjects will receive no AED. Upon completion of the Taper/Washout Period, subjects will begin Treatment Period 2.The procedures and assessments for Treatment Period 1 will be repeated for Treatment Period 2 (with the same duration of treatment).

ELIGIBILITY:
Inclusion Criteria:

* Subjects are between 18 and 55 years of age (inclusive)
* Subjects have a Body Mass Index (BMI) between 18 and 35 kg/m^2 (inclusive)
* Subjects must be in generally good health with no clinically relevant health conditions

Exclusion Criteria:

* Subject has previously been randomized in this study or subject has received LCM or CBZ
* Subjects may not currently be participating in or have participated in the past 30 days in a clinical drug or device study
* Subjects may not have a history of drug or alcohol abuse within the last 2 years
* Subjects may not consume more than 40 g of alcohol per day
* Females who are pregnant or nursing are ineligible; females of childbearing potential must agree to adhere to protocol conception guidelines
* Subjects may not score ≤ 70 on the Peabody Picture Vocabulary Test (PPVT)
* Subjects with a lifetime history of suicide attempt or suicidal ideation in the past 6 months may not participate
* Subjects with a diet that deviates notably from the normal amounts of protein, carbohydrate, and fat, as judged by the investigator are ineligible to participate
* Subjects may not consume more than 600 mg of caffeine/day
* Subjects may not smoke more than 10 cigarettes per day or have done so within 6 months prior to Screening
* Subjects may not have a positive alcohol breath test or urine drug screen at Screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Mean Within-subject Difference In The Overall Neuropsychological Composite Score During Both Treatment Periods | From 6-week Treatment Period 1 to 6-week Treatment Period 2 (Visit 1- Visit 9)
  The overall composite score will be computed as the sum of the individual cognitive test scores from computerized tests and non-computerized neuropsychological tests (including behavioral questionnaires) after transformation to a Z-scores to form an overall composite Z-score. The Z-score will be calculated using the values (mean and standard deviation) from the average of the scores from 3 non-drug conditions (Baseline, first Washout Period, and second Washout Period).

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — 877-822-9493
Locations (2):
- United States (2):
  - 001, Atlanta, Georgia
  - 002, Overland Park, Kansas

REFERENCES:
- [Derived] Meador KJ, Loring DW, Boyd A, Echauz J, LaRoche S, Velez-Ruiz N, Korb P, Byrnes W, Dilley D, Borghs S, De Backer M, Story T, Dedeken P, Webster E. Randomized double-blind comparison of cognitive and EEG effects of lacosamide and carbamazepine. Epilepsy Behav. 2016 Sep;62:267-75. doi: 10.1016/j.yebeh.2016.07.007. Epub 2016 Aug 10. PMID 27517350